CLINICAL TRIAL: NCT01590888
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Tolerability, and Efficacy of PBT2 in Patients With Early to Mid-stage Huntington Disease
Brief Title: Effect of PBT2 in Patients With Early to Mid Stage Huntington Disease
Acronym: Reach2HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prana Biotechnology Limited (Industry)
Responsible Party: Sponsor
Organization: Pranabio (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBT2-203
Record Dates: First submitted 2012-04-18; First posted 2012-05-03 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PBT2 250mg (Experimental)
  Interventions: Drug: PBT2
- PBT2 100mg (Experimental)
  Interventions: Drug: PBT2
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBT2 — 250mg capsules administered orally once per day for 26 weeks
  Arms: PBT2 250mg
Drug: PBT2 — 100mg capsules administered orally once per day for 26 weeks
  Arms: PBT2 100mg
Drug: Placebo — Matching capsules administered orally once per day for 26 weeks
  Arms: Sugar pill

SUMMARY:
Huntington disease (HD) is an inherited neurodegenerative disease which affects over 30,000 people in both the United States and Australia. HD is characterized by brain cell death that usually begins between the ages of 30 to 50, and results in motor, cognitive and behavioral signs and symptoms. While there are medications to help relieve some of the disease symptoms, there is no known treatment to address the cognitive impairment associated with HD.

Normally occurring metals in the brain play a significant role in diseases such as Alzheimer disease and HD. PBT2 is a drug designed to interrupt interactions between these biological metals and target proteins in the brain, to prevent deterioration of brain cells. PBT2, has shown in animal models, and as well as in a small group of patients with Alzheimer's disease, it may improve cognition. There is some indication in animal models of HD, that the drug may improve motor function and control and reduce the amount of brain cell degeneration.

PBT2-203 will evaluate how safe and well tolerated PBT2 is at a dose of 100 mg or 250 mg a day administered as oral daily capsules compared to a placebo over a six month treatment period. The trial will also measure whether there is an effect on cognitive abilities as well as other HD symptoms including motor and overall functioning of individuals with HD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who:

  1. Provide signed informed consent in accordance with local regulations.
  2. Have Huntington disease including clinical features of HD and a CAG repeat number ≥ 36.
  3. Have a Total Functional Capacity between 6 and 13, inclusive.
  4. Have cognitive impairment as demonstrated by a MoCA score of ≥ 12.
  5. Are ≥ 25 years of age.
  6. If taking tetrabenazine, have been on a stable dose for at least 3 months.
  7. If female, are either a) of childbearing potential and compliant in using adequate birth control or b) not of childbearing potential.
  8. If male, is either a) of reproductive potential and compliant in using adequate birth control or b) not of reproductive potential.
  9. Have a study partner who is willing to provide consent and spends on average at least two hours a day for at least four days a week with the patient, is fluent in the English language, and who agrees to attend certain study visits and provide accurate information about the patient.
  10. Are able to swallow oral capsules.
  11. Are fluent in the English language for the administration of rating scales and have sufficient visual, hearing and motor skills to complete procedures.

      Exclusion Criteria:
* Patients who:

  1. Have an allergy to PBT2 or its excipients.
  2. Have other known primary neurodegenerative disorders associated with dementia.
  3. Have known dementia syndromes due to non-primary CNS disease.
  4. Have another condition that in the investigator's judgment is resulting in clinically significant cognitive impairment.
  5. In the opinion of the investigator, have any clinically significant uncontrolled medical or psychiatric illness, including history of seizures.
  6. Have clinically significant cardiovascular, hepatic, renal, pulmonary, metabolic or endocrine disease that, in the opinion of the investigator, would interfere with an individual's participation in the study.
  7. Have a calculated creatinine clearance at Screening of <50mL/min.
  8. Have a history of malignancy diagnosed within 2 years of Screening.
  9. Are pregnant or lactating females.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Dorsey, Principal Investigator — Johns Hopkins University
Locations (19):
- United States (14):
  - University of California San Diego, San Diego, California
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - University of Miami, Miami, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital East, Charlestown, Massachusetts
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Washington University, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
- Australia (5):
  - Westmead Hospital, Sydney, New South Wales
  - Calvary Health Care Bethlehem, Clayton, Victoria
  - University of Melbourne Normanby Unit - St Vincents/St Georges, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Neurodegenerative Disorders Research, Perth, Western Australia

REFERENCES:
- [Background] Lannfelt L, Blennow K, Zetterberg H, Batsman S, Ames D, Harrison J, Masters CL, Targum S, Bush AI, Murdoch R, Wilson J, Ritchie CW; PBT2-201-EURO study group. Safety, efficacy, and biomarker findings of PBT2 in targeting Abeta as a modifying therapy for Alzheimer's disease: a phase IIa, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2008 Sep;7(9):779-86. doi: 10.1016/S1474-4422(08)70167-4. Epub 2008 Jul 30. PMID 18672400
- [Background] Faux NG, Ritchie CW, Gunn A, Rembach A, Tsatsanis A, Bedo J, Harrison J, Lannfelt L, Blennow K, Zetterberg H, Ingelsson M, Masters CL, Tanzi RE, Cummings JL, Herd CM, Bush AI. PBT2 rapidly improves cognition in Alzheimer's Disease: additional phase II analyses. J Alzheimers Dis. 2010;20(2):509-16. doi: 10.3233/JAD-2010-1390. PMID 20164561
- [Derived] Huntington Study Group Reach2HD Investigators. Safety, tolerability, and efficacy of PBT2 in Huntington's disease: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2015 Jan;14(1):39-47. doi: 10.1016/S1474-4422(14)70262-5. Epub 2014 Nov 14. PMID 25467848
- [Derived] Cherny RA, Ayton S, Finkelstein DI, Bush AI, McColl G, Massa SM. PBT2 Reduces Toxicity in a C. elegans Model of polyQ Aggregation and Extends Lifespan, Reduces Striatal Atrophy and Improves Motor Performance in the R6/2 Mouse Model of Huntington's Disease. J Huntingtons Dis. 2012;1(2):211-9. doi: 10.3233/JHD-120029. PMID 25063332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty sites were initiated for the study, with participants enrolled at 14 sites in the US and 5 sites in Australia.
Period: Overall Study
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Started | 36 | 38 | 35
Completed | 32 | 38 | 34
Not Completed | 4 | 0 | 1
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill | Total
Number analyzed (Participants) | 36 | 38 | 35 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.4) | 54.1 (12.1) | 51.2 (10.4) | 51.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 19 | 55
  Male | 19 | 19 | 16 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 34 | 38 | 35 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 35 | 38 | 35 | 108
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 25 | 79
  Australia | 10 | 10 | 10 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.51 (4.89) | 25.40 (4.53) | 27.09 (6.03) | 25.98 (5.18)
Total Function Capacity [Mean (Standard Deviation); unit: units on a scale] — Total function capacity (TFC) is a scale measuring the participants capacity to perform 5 areas - their capacity to work, capacity to handle financial affairs, capacity to manage domestic responsibilities, capacity to perform activities of daily living and level of care required (home or care facility). The scale used is a TOTAL of each of the 5 areas, which range from 0 (unable to perform or require full care) to either 2 or 3 (normal, no assistance required). The TFC can scored from 0 to 13. The lower the score, the more severe the disease state of Huntington disease is.
  units on a scale | 9.1 (2.2) | 9.3 (2.3) | 9.3 (1.6) | 9.2 (2.0)
CAG Larger Allele Repeat Length [Mean (Standard Deviation); unit: CAG repeats] — Huntington disease (HD) is a dominant genetic disorder. Mutations in the HTT gene cause HD. The HTT mutation involves a DNA segment known as a Cytosine, Adenine and Guanine (CAG) trinucleotide repeat, a series of three DNA building blocks. Normally, the CAG segment is repeated 10 to 35 times within the gene. In people with HD, the CAG segment is repeated more than 36 times with higher repeat numbers normally indicating earlier onset of the disease and increased severity of symptoms.
  CAG repeats | 44.4 (4.6) | 43.2 (2.8) | 44.1 (3.9) | 43.9 (3.8)
CAG Smaller Allele Repeat Length [Mean (Standard Deviation); unit: CAG repeats] — Huntington disease (HD) is a dominant genetic disorder. Mutations in the HTT gene cause HD. The HTT mutation involves a DNA segment known as a Cytosine, Adenine and Guanine (CAG) trinucleotide repeat, a series of three DNA building blocks. Normally, the CAG segment is repeated 10 to 35 times within the gene. In people with HD, the CAG segment is repeated more than 36 times with higher repeat numbers normally indicating earlier onset of the disease and increased severity of symptoms.
  HD is a dominant genetic disorder.
  CAG repeats | 18.8 (4.4) | 18.5 (3.0) | 20.0 (4.8) | 19.1 (4.1)
Disease Burden [Mean (Standard Deviation); unit: CAG repeats*years] — Disease burden in patients with Huntington disease is calculated by (CAG repeat length - 35) x Age at Baseline, with the higher score indicating a greater Disease Burden for a patient.
  CAG repeats*years | 411.68 (104.96) | 392.54 (96.10) | 410.07 (110.02) | 404.49 (103.06)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of PBT2 in Patients With HD
Description: As measured by the total number of participants in each dose group who reported at least one adverse events during the study,
Time Frame: Baseline to 26 weeks
Population: Safety population as defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 36 | 38 | 35
participants | 32 | 30 | 28

2. Secondary Outcome: Change From Baseline in Cognitive Test Battery - Composite z Scores
Description: Cognition composite z-scores were calculated for each participant. The composite scores were defined as the mean of the individual z-scores for the various cognition assessments. The Main Composite z-score was calculated for Category Fluency Test, Trail Making Test Part B, Map Search, Symbol Digit Modalities Test and Stroop Word Reading Test. The Exploratory Composite z-score was calculated for Category Fluency Test, Trail Making Test Part B, Map Search, Symbol Digit Modalities Test, Stroop Word Reading Test and Speeded Tapping test. The Executive Function Composite z-score was calculated from Category Fluency Test and Trail Making Test Part B. There is no unit of measure for the z score as it is the pure number calculated from the SD from the mean. A higher z score indicates an improvement.
Time Frame: Baseline to 26 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 32 | 38 | 34
z score
  Main Composite z-score | 0.0592 (0.2670) | -0.0413 (0.3170) | -0.0194 (0.2374)
  Exploratory Composite z-score | 0.0530 (0.2568) | -0.0287 (0.3349) | -0.0144 (0.2331)
  Executive Function z-score | 0.2274 (0.4288) | -0.1026 (0.4771) | 0.0553 (0.3385)

3. Secondary Outcome: Change From Baseline in Motor Function
Description: Total motor score calculated from the Unified Huntington Disease Rating Scale - Motor Function. The motor section of the UHDRS assesses motor features of HD with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural stability. The total motor impairment scores is the sum of all the individual motor ratings, with higher scores indicating more severe motor impairment than lower scores. A maximum score of 60 is possible (range 0-60).
Time Frame: Baseline to 26 weeks
Population: Intent to Treat population analysed, and defined as all participants who received at least one dose of study and underwent at least one post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 34 | 38 | 35
units on a scale | -0.7 (7.6) | 1.3 (9.0) | -1.3 (7.3)

4. Secondary Outcome: Change From Baseline in Functional Abilities
Description: Total Functional Capacity (TFC) assessment was based on an individual's ability to perform common daily tasks. TFC score range was 0 to 13.
  Higher scores on the function scales indicate better functioning than lower scores.
Time Frame: Baseline to 26 weeks
Population: Intent to Treat Population analysed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 34 | 38 | 35
units on a scale | 1.1 (1.0) | 1.3 (1.0) | 1.3 (0.9)

5. Secondary Outcome: Change From Baseline in Behaviour
Description: Total Behavioural score from the Unified Huntington Disease Rating Scale. The behavioural assessment measures the frequency and severity of symptoms related to affect, thought content and coping styles. The total behaviour score is the sum of all responses, with scale range of 0 to 8. Higher scores on the behaviour assessments indicate more severe disturbance than lower scores.
Time Frame: Baseline to 26 weeks
Population: Intent to Treat population analysed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 34 | 38 | 35
units on a scale | -2.3 (9.2) | 3.0 (15.9) | 0.7 (13.0)

6. Secondary Outcome: Change From Baseline in Investigator Global Assessments by Efficacy Index
Description: Global function was assessed by the Investigator using the clinical global impression (CGI) scale which included assessing the severity of illness and global improvement and calculating the efficacy index for each participant. The efficacy index aims to relate therapeutic effects to reported side effects as assessed by the Investigator (range from 0 [marked improvement and no side effects] to 4 [unchanged or worse] and side effects outweigh therapeutic effects) and is calculated for each participant by dividing the therapeutic effect score by the side effects score. An improvement is reflected by CGI scale Efficacy Index values >1.
Time Frame: Baseline to 26 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 32 | 38 | 34
ratio | 1.313 (0.592) | 1.276 (0.654) | 1.176 (0.459)

7. Secondary Outcome: Change From Baseline in Blood Biomarkers
Description: Biomarkers assessed primarily with mutant huntingtin protein, normalised to lysate protein concentrations, as a change from baseline.
Time Frame: Baseline to 26 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 32 | 38 | 34
ratio | 1.97 (24.39) | 0.14 (4.70) | -1.72 (9.72)

8. Secondary Outcome: Change From Baseline in Brain Function (MRI)
Description: Measure of whole brain iron concentrations.
Time Frame: Baseline to 26 weeks
Population: ITT population. MRI was performed at one site only, resulting in a subset of participants available for analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 2 | 1 | 2
mm^3 | 0.0029 (0.0043) | 0.0067 (NA) — Not applicable with an n equalling 1. | 0.0098 (0.0115)

9. Secondary Outcome: Change From Baseline in Blood Biomarkers
Description: Biomarkers assessed primarily with soluble huntingtin protein, normalised to lysate protein concentrations, as a change from baseline.
Time Frame: Baseline to 26 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 23 | 27 | 28
mg/mL | -3.18 (8.23) | -2.09 (5.44) | -3.07 (5.98)

10. Secondary Outcome: Change From Baseline in Blood Biomarkers - Selenium
Description: Biomarkers assessed primarily with plasma selenium as a change from baseline.
Time Frame: Baseline to 26 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 32 | 35 | 33
ug/L | 1.3 (28.1) | -6.3 (18.2) | 2.0 (20.5)

11. Secondary Outcome: Change From Baseline in Urine Biomarkers
Description: Biomarkers assessed primarily with 8-hydroxy-2'-deoxyguanosine, normalised to creatinine concentrations, as a change from baseline.
Time Frame: Baseline to 26 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 30 | 38 | 33
ng/mL | -0.4258 (1.3383) | 0.0832 (2.0456) | 35.5302 (208.5614)

12. Secondary Outcome: Change From Baseline in Brain Function (MRI)
Description: Measure of the structural brain volume as assessed by the left caudate volume.
Time Frame: Baseline to 26 weeks
Population: ITT population. MRI was performed at one site only, resulting in a subset of participants available for analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 2 | 2 | 2
mm^3 | 50.0 (70.7) | 27.5 (94.0) | -170.5 (67.2)

13. Secondary Outcome: Change From Baseline in Cognitive Test Battery - TMT Part B
Description: Trail Making Test Part B was assessed by the number of seconds to complete the test (from 0 to 240 seconds).
  The Trails Making Test Part B actual change from baseline at Week 26 was analysed.
Time Frame: Baseline to 26 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Number analyzed (Participants) | 32 | 38 | 34
seconds | -6.3 (30.0) | 12.8 (43.3) | 8.9 (28.7)

ADVERSE EVENTS:
Time Frame: Reported AEs from time of consent to end of study (Week 30 or 4 weeks post cessation of study drug).
Arm/Group | PBT2 250mg | PBT2 100mg | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 5/36 | 2/38 | 1/35
Other Adverse Events (participants affected / at risk) | 3/36 | 3/38 | 2/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBT2 250mg (N=36) | PBT2 100mg (N=38) | Sugar Pill (N=35)
Psychotic Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening of Huntington Disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stabilisation of Huntington Disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBT2 250mg (N=36) | PBT2 100mg (N=38) | Sugar Pill (N=35)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Huntington disease (Congenital, familial and genetic disorders) | 1 (1) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Muscolskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less